CLINICAL TRIAL: NCT03203551
Title: Clinical and Laboratorial Evaluation of the Effect of Sodium Hypochlorite, Chloramine T and Ricinus Communis Solutions in Candida Species Identified in the Biofilm of Total Prostheses and Palate of Total Edentulous Individuals.
Brief Title: Clinical and Laboratorial Evaluation of the Desinfection Solutions in Candida Species From Total Prostheses and Palate of Total Edentulous.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Cláudia Helena Lovato da Silva, Principal Investigator and Clinical Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FORP/USP
Record Dates: First submitted 2017-06-23; First posted 2017-06-29 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Candidiasis; Biofilms; Candida Infection
Keywords: Dentures; Biofilms; Disinfection; Candidiasis; Candida
MeSH Terms: conditions — Candidiasis; Torulopsis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- C; Control; Saline solution (Placebo Comparator): Disinfection protocol:
  * brushing the palate (3 times a day/ 2 minutes);
  * brushing the total prostheses with neutral liquid soap (3 times a day/ 3 minutes);
  * immersing the total prostheses in Saline solution (once a day/ 20 minutes) before the last brushing of the day;
  * the prostheses must be conditioned in a vessel with water during the whole night period.
  Periods of analysis (Baseline, 7 and 37 days):
  * the prostheses will be evidenced and photographed.
  * the biofilm present on the inner surface of the prostheses will be collected;
  * photographe of the participants' palate;
  * collected the palate biofilm.
  Interventions: Other: Disinfection Protocol
- HS0.25%; 0.25% Sodium Hypochlorite (Experimental): Disinfection protocol:
  * brushing the palate (3 times a day/ 2 minutes);
  * brushing the total prostheses with neutral liquid soap (3 times a day/ 3 minutes);
  * immersing the total prostheses in 0.25% Sodium Hypochlorite (once a day/ 20 minutes) before the last brushing of the day;
  * the prostheses must be conditioned in a vessel with water during the whole night period.
  Periods of analysis (Baseline, 7 and 37 days):
  * the prostheses will be evidenced and photographed.
  * the biofilm present on the inner surface of the prostheses will be collected;
  * photographe of the participants' palate;
  * collected the palate biofilm.
  Interventions: Other: Disinfection Protocol
- RC10%; 10% Ricinus communis (Experimental): Disinfection protocol:
  * brushing the palate (3 times a day/ 2 minutes);
  * brushing the total prostheses with neutral liquid soap (3 times a day/ 3 minutes);
  * immersing the total prostheses in 10% Ricinus communis (once a day/ 20 minutes) before the last brushing of the day;
  * the prostheses must be conditioned in a vessel with water during the whole night period.
  Periods of analysis (Baseline, 7 and 37 days):
  * the prostheses will be evidenced and photographed.
  * the biofilm present on the inner surface of the prostheses will be collected;
  * photographe of the participants' palate;
  * collected the palate biofilm.
  Interventions: Other: Disinfection Protocol
- CT0.5%; 0.5% Chloramine T (Experimental): Disinfection protocol:
  * brushing the palate (3 times a day/ 2 minutes);
  * brushing the total prostheses with neutral liquid soap (3 times a day/ 3 minutes);
  * immersing the total prostheses in 0.5% Choramine T (once a day/ 20 minutes) before the last brushing of the day;
  * the prostheses must be conditioned in a vessel with water during the whole night period.
  Periods of analysis (Baseline, 7 and 37 days):
  * the prostheses will be evidenced and photographed.
  * the biofilm present on the inner surface of the prostheses will be collected;
  * photographe of the participants' palate;
  * collected the palate biofilm.
  Interventions: Other: Disinfection Protocol

INTERVENTIONS:
Other: Disinfection Protocol — The participants assigned to this group carried out the disinfection protocol that recommended brushing the palate (3 times a day), brushing the total prosthesis with neutral liquid soap (3 times a day) and immersing in different desinfection solutions (once a day/ 20 minutes)
  Other Names: Denture Hygiene Protocol

SUMMARY:
This clinical study identified the Candida species from the palate and complete dentures of edentulous individuals with prostheses-related stomatitis (PRS) and evaluated the effect of disinfectant solutions for denture hygiene on Candida spp. Sixty participants were randomly assigned in 04 parallel groups (n = 15); They were oriented to brush their prostheses and the palate 3 times a day and immerse them in saline solution (C-control), 0.25% Sodium hypochlorite (HS0.25%), 10% Ricinus communis (RC10%) or 0.5% Chloramine T (CT 0.5%) for 20 minutes. Biofilm samples were collected from the prostheses and palate in the baseline, after 7 and 37 days of use of the solutions and seeded in CHROMagar Candida medium. After incubation period, the presumptive identification, incidence verification and quantification of Candida species growth (CFU count) were performed. To quantify biofilm with software ImageTool 3.0, the inner surface was disclosed (1% neutral red) and photographed at the end of each period. The Candidiasis remission was assessed by scores before and after the use of solutions by palate's phographs. Descriptive analyzes were used for the identification and incidence of Candida spp. Kruskal-Wallis and Friedman tests, with stepwise step-down post-test for cell growth; ANOVA and Tukey for biofilm removal; Frequency of scores for evolution of inflammation. Level of significance was 95%. The most incident species were C. albicans, followed by C. tropicalis, C. glabrata and C. krusei. HS 0.25% reduced the incidence of the three species on the prostheses and palate in the periods of 7 and 37 days; CT 0.5% promoted reduction of Candida spp. only in dentures. R. communis decreased the incidence of C. tropicalis in both collection sites. For CFU counts, HS 0.25% and CT 0.5% caused significant reduction. For biofilm removal, HS0.25% was the most effective (9.75 ± 12.6) and RC10% (15.92 ± 14.8) intermediate. All groups decreased protheses-related stomatitis. HS0.25% has potential for clinical use as total denture disinfectants. RC10% and CT0.5% require further studies to be indicated as alternative solutions.

ELIGIBILITY:
Inclusion criteria:

* providing consent prior to participation in the study;
* being at least 18 years of age;
* maxillary complete conventional denture in good state and 1 year of use;
* dentures with biofilm in a internal surface;
* moderate to severe signs of Candidiasis.

Exclusion criteria:

* presence oral mucosal lesions apart from Candidiasis;
* systemic or local conditions which predispose to Candida spp. infection;
* history of chemotherapy/ radiotherapy;
* having taken or used antibiotics, steroidal agents, or antifungal agents in the three months prior to the study;
* being scheduled to replace existing dentures with new ones during the period of the trial;
* dentures with adaptation or retention problems;
* already using palatal brushing or disinfectant solutions as a routine oral hygiene.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation of the Candida species identified in the biofilm of total prostheses and palate of total edentulous individuals. | Baseline (without disinfection procedures)
  Biofilm samples were collected from the prosthesis and palate in the baseline and seeded in CHROMagar Candida medium. After incubation period, the presumptive identification, incidence verification and quantification of Candida species growth (CFU count) were performed. The inner surface of the denture was disclosed (1% neutral red) and photographed at the end to quantify the biofilm with the software ImageTool 3.0. The palate with Candidiasis was photographed and assessed by scores.

SECONDARY OUTCOMES:
Clinical evaluation of the effect of Sodium hypochlorite, Chloramine T and Ricinus communis solutions after 7 days of use in Candida species identified in the biofilm of total prostheses and palate of total edentulous individuals. | 7 days of disinfection
  Biofilm samples were collected from the prostheses and palate after 7 days of use of the solutions and seeded in CHROMagar Candida medium. After incubation period, the presumptive identification, incidence verification and quantification of Candida species growth (CFU count) were performed. To quantify the denture biofilm with software ImageTool 3.0, the inner surface of the denture was disclosed (1% neutral red) and photographed at the end of 7 days. The Candidiasis remission was photographed and assessed by scores after 7 days of use solutions.
Clinical evaluation of the effect of Sodium hypochlorite, Chloramine T and Ricinus communis solutions after 37 days of use in Candida species identified in the biofilm of total prostheses and palate of total edentulous individuals. | 37 days of disinfection
  Biofilm samples were collected from the prostheses and palate after 37 days of use of the solutions and seeded in CHROMagar Candida medium. After incubation period, the presumptive identification, incidence verification and quantification of Candida species growth (CFU count) were performed. To quantify the denture biofilm with software ImageTool 3.0, the inner surface of the denture was disclosed (1% neutral red) and photographed at the end of 37 days. The Candidiasis remission was photographed and assessed by scores after 37 days of use solutions.

IPD SHARING:
Plan to Share IPD: No